CLINICAL TRIAL: NCT02511158
Title: Prospective Follow-up Study of Patients Undergoing Knee Ligament Surgery
Brief Title: French Prospective Anterior Cruciate Ligament Reconstruction Cohort Study (FAST)
Acronym: FAST
Status: Recruiting | Type: Observational
Sponsor: Fonds de Dotation pour la Recherche Clinique en Orthopédie et Pathologie du Sport (Other)
Responsible Party: Principal Investigator, Shahnaz Klouche, Physician responsible of clinical research, Fonds de Dotation pour la Recherche Clinique en Orthopédie et Pathologie du Sport
Other Study IDs: CMC2012
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Rupture of Anterior Cruciate Ligament; Osteoarthritis
Keywords: Anterior Cruciate Ligament, Posterior Cruciate Ligament, Medial Collateral Ligament, Lateral Collateral Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ligament of the knee reconstruction — Reconstruction of ligaments of the knee by autografts

SUMMARY:
In this study we will examine patients who have undergone anterior cruciate and/or posterior cruciate ligament and/or multi ligaments reconstruction to determine the rate of re-injury, contralateral tear and functional outcomes at least two years after surgery.

DETAILED DESCRIPTION:
The purpose of this study is to identify the rate of re tear two year after ligament reconstruction of the knee. The second objective is to assess the osteoarthritis of the knee at 20 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* One ligament or multi-ligaments tear of the knee
* Surgery reconstruction with any technique

Exclusion Criteria:

* Patient refusal

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants enrolled in the FAST cohort by one of four surgeons and meeting eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2012-09; Primary Completion 2032-09 (Estimated); Study Completion 2052-09 (Estimated)

PRIMARY OUTCOMES:
Number of re-tear | 2 years

SECONDARY OUTCOMES:
International Knee Documentation Committee score | 2 years
Lyshom score | 2 years
Tegner score | 2 years
Knee injury and Osteoarthritis Outcome Score | 2 years
joint line space measurement on comparative standard radiograph at 30 degree of flexion before surgery and at the final follow-up (Schuss view) | 20 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Médico-Chirurgical Paris V (CMCV), Paris, France

REFERENCES:
- [Result] Lefevre N, Klouche S, de Pamphilis O, Devaux C, Herman S, Bohu Y. Postoperative discomfort after outpatient anterior cruciate ligament reconstruction: a prospective comparative study. Orthop Traumatol Surg Res. 2015 Apr;101(2):163-6. doi: 10.1016/j.otsr.2014.07.036. Epub 2015 Feb 7. PMID 25666422
- [Result] Lefevre N, Bohu Y, de Pamphilis O, Klouche S, Devaux C, Herman S. Outpatient surgery feasibility in anterior cruciate ligament reconstruction: a prospective comparative assessment. Orthop Traumatol Surg Res. 2014 Sep;100(5):521-6. doi: 10.1016/j.otsr.2014.03.024. Epub 2014 Jul 28. PMID 25082774
- [Result] Bohu Y, Klouche S, Lefevre N, Webster K, Herman S. Translation, cross-cultural adaptation and validation of the French version of the Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) scale. Knee Surg Sports Traumatol Arthrosc. 2015 Apr;23(4):1192-6. doi: 10.1007/s00167-014-2942-4. Epub 2014 Mar 28. PMID 24676789
- [Result] Lefevre N, Naouri JF, Bohu Y, Klouche S, Herman S. Sensitivity and specificity of bell-hammer tear as an indirect sign of partial anterior cruciate ligament rupture on magnetic resonance imaging. Knee Surg Sports Traumatol Arthrosc. 2014 May;22(5):1112-8. doi: 10.1007/s00167-013-2511-2. Epub 2013 Apr 21. PMID 23604176
- [Result] Lefevre N, Bohu Y, Naouri JF, Klouche S, Herman S. Validity of GNRB(R) arthrometer compared to Telos in the assessment of partial anterior cruciate ligament tears. Knee Surg Sports Traumatol Arthrosc. 2014 Feb;22(2):285-90. doi: 10.1007/s00167-013-2384-4. Epub 2013 Jan 22. PMID 23338663
- [Result] Sadeqi M, Klouche S, Bohu Y, Herman S, Lefevre N, Gerometta A. Progression of the Psychological ACL-RSI Score and Return to Sport After Anterior Cruciate Ligament Reconstruction: A Prospective 2-Year Follow-up Study From the French Prospective Anterior Cruciate Ligament Reconstruction Cohort Study (FAST). Orthop J Sports Med. 2018 Dec 17;6(12):2325967118812819. doi: 10.1177/2325967118812819. eCollection 2018 Dec. PMID 30574516
- [Result] Bohu Y, Klouche S, Herman S, de Pamphilis O, Gerometta A, Lefevre N. Professional Athletes Are Not at a Higher Risk of Infections After Anterior Cruciate Ligament Reconstruction: Incidence of Septic Arthritis, Additional Costs, and Clinical Outcomes From the French Prospective Anterior Cruciate Ligament Study (FAST) Cohort. Am J Sports Med. 2019 Jan;47(1):104-111. doi: 10.1177/0363546518810527. Epub 2018 Nov 27. PMID 30481480
- [Result] Raoul T, Klouche S, Guerrier B, El-Hariri B, Herman S, Gerometta A, Lefevre N, Bohu Y. Are athletes able to resume sport at six-month mean follow-up after anterior cruciate ligament reconstruction? Prospective functional and psychological assessment from the French Anterior Cruciate Ligament Study (FAST) cohort. Knee. 2019 Jan;26(1):155-164. doi: 10.1016/j.knee.2018.11.006. Epub 2018 Nov 22. PMID 30473373
- [Result] Lefevre N, Klouche S, de Pamphilis O, Herman S, Gerometta A, Bohu Y. Peri-articular local infiltration analgesia versus femoral nerve block for postoperative pain control following anterior cruciate ligament reconstruction: Prospective, comparative, non-inferiority study. Orthop Traumatol Surg Res. 2016 Nov;102(7):873-877. doi: 10.1016/j.otsr.2016.07.011. Epub 2016 Oct 4. PMID 27720193
- [Result] Lefevre N, Klouche S, Mirouse G, Herman S, Gerometta A, Bohu Y. Return to Sport After Primary and Revision Anterior Cruciate Ligament Reconstruction: A Prospective Comparative Study of 552 Patients From the FAST Cohort. Am J Sports Med. 2017 Jan;45(1):34-41. doi: 10.1177/0363546516660075. Epub 2016 Aug 20. PMID 27530413
- [Derived] Moussa MK, Lefevre N, Valentin E, Coughlan A, Zgolli A, Gerometta A, Meyer A, Hardy A. Impact of Lateral Extra-Articular Procedure Augmentation on Rerupture Risk and Tegner Activity Scale Outcomes in Adolescent Anterior Cruciate Ligament: A Matched Comparative Study With a Minimum 2-Year Follow-up. Am J Sports Med. 2024 Mar;52(4):892-901. doi: 10.1177/03635465231223703. Epub 2024 Feb 9. PMID 38333967
- [Derived] Bohu Y, Klouche S, Sezer HB, Herman S, Grimaud O, Gerometta A, Meyer A, Lefevre N. Vancomycin-soaked autografts during ACL reconstruction reduce the risk of post-operative infection without affecting return to sport or knee function. Knee Surg Sports Traumatol Arthrosc. 2020 Aug;28(8):2578-2585. doi: 10.1007/s00167-020-05879-9. Epub 2020 Feb 5. PMID 32025764